CLINICAL TRIAL: NCT00529698
Title: A Phase I Safety and Immunogenicity Trial of Recombinant HIV-1 Tat Protein in HIV-1 Uninfected Adult Volunteers
Brief Title: Phase I Safety and Immunogenicity Preventative Vaccine Trial Based on Recombinant Tat Protein
Acronym: ISSP-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Responsible Party: Barbara Ensoli, MD, Phd, Istituto Superiore di Sanita
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ISSP-001
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: HIV; Tat protein; Preventative vaccine; Healthy volunteers; HIV-1/2 uninfected; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Subjects were immunized subcutaneously with Tat, 3 dosage groups (7.5, 15 or 30 micrograms), in association with Alum as adjuvant, or with Saline + Alum, as placebo.
  Interventions: Biological: Biologically active recombinant Tat protein
- B (Other): Subjects were immunized intradermally with Tat, 3 dosage groups (7.5, 15 or 30 micrograms), or with Saline, as placebo.
  Interventions: Biological: Biologically active recombinant Tat protein

INTERVENTIONS:
Biological: Biologically active recombinant Tat protein

SUMMARY:
This Phase I study is directed at evaluating the safety profile (as a primary end-point) and the immunogenicity (as a secondary end-point) of the recombinant HIV-1 Tat vaccine in healthy, immunologically competent adult subjects without identifiable risk of HIV-1 infection.

DETAILED DESCRIPTION:
The development of a vaccine against HIV/AIDS has been primary focused on the structural proteins (Env, Gag) of HIV-1 with the aim of inducing sterilizing immunity by blocking virus entry. Alternative approaches are focused on new vaccine strategies aimed at modifying the virus-host dynamic favouring the establishment of a long-term non-progressing disease status. Such strategies target regulatory proteins that are the first to be expressed after infection and are essential for viral replication, infectivity and pathogenesis. Thus, this approach may be effective for both preventive and therapeutic vaccination strategies.

Being a very early viral regulatory protein necessary for viral gene expression, cell-to-cell virus transmission and disease progression, Tat represents a key target protein for the host immune response and an optimal candidate for such a vaccination strategy.

Preclinical studies demonstrated that vaccination with a biologically active Tat protein is safe, elicits a broad and specific immune response and induces a long-term protection against infection. Cross-sectional and longitudinal studies in natural infection suggest that the presence of an anti-Tat humoral immune response correlates with asymptomatic infection and with a slower disease progression while the presence of CD8+ T cell responses to Tat correlate with early virus control both in humans and monkeys. Since the immunogenic regions of Tat are well conserved among the HIV-1 M group, a vaccine based on Tat may be used in different geographic areas of the world.

The subjects were stratified in two Arms according to the administration route to receive 5 intradermal or subcutaneous immunizations at 4 weeks intervals.

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy test for women of childbearing potential within 3 days prior to baseline evaluation and use of an acceptable means of contraception (condom, hormonal or mechanical method) for one month prior to immunization and for all the duration of the study;
* Complete blood count and differential defined as:
* Hematocrit >=30% for women, >= 38% for men
* Hemoglobin >= 9.5 g/dL
* White cell counts >= 4,000 and <= 9,500 cells/mm3
* Total lymphocyte count >=1000 cells/mm3
* CD4+ T cell count > 500 cells/microL based on 2 separate determinations (Hannet, 1992)
* Platelets (100,000-550,000/ mm3)
* Differential within institutional normal limits or approval of site physician;
* Normal ALT (as defined by the range of the clinical site laboratory) and Creatinine (< 1.6 mg/dl);
* Normal urine dipstick with esterase and nitrite;
* Normal thyroid function;
* Negative ELISA for HIV-1/HIV-2 and HIV-1 viral load (plasma viremia) < 50 copies/mL within 1 month of immunization;
* Availability for follow-up for planned duration of at least 12 months and willing to have further brief evaluations at 24 and 36 months;
* Signed informed consent.

Exclusion Criteria:

* Identifiable high-risk behavior for HIV-1 infection, including a history of injection drug use within 12 months prior to enrollment or higher-risk sexual behavior;
* History of neoplastic diseases, encephalopathy, neuropathy or unstable CNS pathology, immunodeficiency, autoimmune disease, angina or cardiac arrhythmias, or any other clinically significant medical problems;
* Chest radiography showing evidence of active or acute cardiac or pulmonary disease;
* History of anaphylaxis or serious adverse reactions to vaccines as well as serum IgE levels exceeding 1000 U.I./ml;
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g. Steven-Johnson syndrome, bronchospasm, or hypotension);
* Active syphilis [NOTE. If the serology is documented to be a false positive or due to an adequately treated infection, the volunteer is eligible];
* Active tuberculosis [NOTE: Volunteers with a positive PPD and a normal chest X-ray showing no evidence of TB and not requiring isoniazid (INH) therapy are eligible];
* Medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol. Specifically excluded are persons with psychotic disorders, major affective disorders, suicidal ideation;
* Current use of psychotropic drugs;
* Participation in another experimental protocol within six months prior to pre-study screening;
* Current or prior therapy with immunomodulators or immunosuppressive drugs and anticoagulant drugs within 30 days prior to study medication administration;
* Any unstable cardiovascular disease (e.g. unstable hypersensitive disease needing modification or introduction of an anti-hypersensitive treatment);
* Live attenuated vaccines within 60 days of study [NOTE: Medically indicated sub-unit or killed vaccines (e.g., influenza, pneumococcal, hepatitis A and B) are not exclusionary, but should be given at least 4 weeks away from HIV immunizations];
* Use of investigational agents within 90 days prior to study;
* Receipt of blood products or immunoglobulin in the past 6 months;
* Prior receipt of HIV-1 vaccine in a previous HIV vaccine trial;
* Positivity for HBV antigens (HBs Ag, HBe Ag), and HCV, HTLV-I and HTLV-II antibodies;
* Pregnant or lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Assessment of safety includes clinical observation and monitoring of haematological, biochemical, virological and immunological parameters. Safety is evaluated by monitoring of volunteers for local and systemic adverse reactions during the trial.

SECONDARY OUTCOMES:
To qualify Tat protein as immunogenic, volunteers are monitored for anti-Tat specific antibodies, anti-Tat proliferative response and in vitro gamma-IFN and IL-4 (or IL-10) production in response to Tat (Elispot).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ensoli, MD, PhD, Study Director — National AIDS Center, Istituto Superiore di Sanita, Rome, Italy
Locations (4):
- Italy (4):
  - San Raffaele Hospital, Milan
  - Hospital Spallanzani, Rome
  - San Gallicano Hospital, Rome
  - University of Rome "La Sapienza", Rome

REFERENCES:
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Cafaro A, Caputo A, Fracasso C, Maggiorella MT, Goletti D, Baroncelli S, Pace M, Sernicola L, Koanga-Mogtomo ML, Betti M, Borsetti A, Belli R, Akerblom L, Corrias F, Butto S, Heeney J, Verani P, Titti F, Ensoli B. Control of SHIV-89.6P-infection of cynomolgus monkeys by HIV-1 Tat protein vaccine. Nat Med. 1999 Jun;5(6):643-50. doi: 10.1038/9488. PMID 10371502
- [Background] Cafaro A, Caputo A, Maggiorella MT, Baroncelli S, Fracasso C, Pace M, Borsetti A, Sernicola L, Negri DR, Ten Haaft P, Betti M, Michelini Z, Macchia I, Fanales-Belasio E, Belli R, Corrias F, Butto S, Verani P, Titti F, Ensoli B. SHIV89.6P pathogenicity in cynomolgus monkeys and control of viral replication and disease onset by human immunodeficiency virus type 1 Tat vaccine. J Med Primatol. 2000 Aug;29(3-4):193-208. doi: 10.1034/j.1600-0684.2000.290313.x. PMID 11085582
- [Background] Butto S, Fiorelli V, Tripiciano A, Ruiz-Alvarez MJ, Scoglio A, Ensoli F, Ciccozzi M, Collacchi B, Sabbatucci M, Cafaro A, Guzman CA, Borsetti A, Caputo A, Vardas E, Colvin M, Lukwiya M, Rezza G, Ensoli B; Tat Multicentric Study Group. Sequence conservation and antibody cross-recognition of clade B human immunodeficiency virus (HIV) type 1 Tat protein in HIV-1-infected Italians, Ugandans, and South Africans. J Infect Dis. 2003 Oct 15;188(8):1171-80. doi: 10.1086/378412. Epub 2003 Sep 30. PMID 14551888
- [Derived] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- See also: Related Info — http://www.iss.it